CLINICAL TRIAL: NCT03630003
Title: Manually Operated Communication System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: J. Matthias Walz (Other)
Collaborators: Brown University (Other)
Responsible Party: Sponsor-Investigator, J. Matthias Walz, Professor and Interim Chair, Dept of Anesthesiology and Perioperative Medicine, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: H00015391
Record Dates: First submitted 2018-08-03; First posted 2018-08-14 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Communication; Ventilation Therapy; Complications
Keywords: ICU; critical care; alternative communication; augmentative communication
MeSH Terms: conditions — Communication | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Use of MOCS with post-use interview (Experimental): The patients in this arm will be asked to utilize the Manually Operated Communication System (MOCS) device and will then be asked to provide feedback on their experiences.
  Subjects will be asked to complete up to 3 sessions using the device. Each session is expected to last between 10 and 30 minutes. If the subject is interested in continuing, the session may last up to one hour.
  The study team will perform post-study interviews with each subject to ask about their experience with MOCS. The data collection forms will be filled out during the session by a member of the research team.
  Interventions: Device: MOCS; Other: Post-use interview

INTERVENTIONS:
Device: MOCS — The device consists of a tablet computer that can produce visual and auditory components designed to improve subject knowledge about setting and communication, mounted on a table or at the side of the bed in a place that is visible to the subject.
  The Arduino will be connected to switches/buttons and implemented in a 3D-printed platform.
  Other Names: Manually Operated Communication System
Other: Post-use interview — The Study team conducts an interview with participants to evaluate their experience with use of the MOCS device.
  Other Names: Interview

SUMMARY:
The objective of this study is to gather initial information about the testing of a novel manual communication system - which is currently called MOCS, for Manually Operated Communicated System - for mechanically ventilated Intensive Care Unit (ICU) subjects. This study is not hypothesis based; the goal is to gather data about which interaction modes and teaching approaches of MOCS are most intuitive for subjects and caregivers.

DETAILED DESCRIPTION:
Intensive Care Unit (ICU) admissions constitute a major part of hospital activity and resource allocation, and the number of patient days in ICUs and on mechanical ventilation is increasing. More than 5 million patients are admitted to an ICU annually in the United States, and approximately 55,000 critically ill patients are cared for each day. The most common cause for admission is respiratory insufficiency or failure; a study of data from 2005-2007 estimated that nearly 40 percent of ICU patients require mechanical ventilation.

Patients experience frequent emotional and psychiatric complications from ICU stays, including depression, anxiety, and post-traumatic stress disorder. One 2011 study found a prevalence of "clinically significant" depressive symptoms ranging from 17 percent to 43 percent among post-ICU patients. In 2013, it was reported that up to 50 percent of patients experience general anxiety symptoms one year after discharge, a rate much higher than in the broader US population.

Patients who temporarily lose the ability to speak report a high level of frustration. A study of 127 patients reported that, "two stressors, being intubated and not being able to talk, were significantly more stressful… than all the other stressors. The mean stressfulness score for [25] other stressors was between no distress and mild distress." Improving subject communication with ICU care team will likely require better technological interventions, and current best practice for assessing the optimal patient communication method is dependent on the evaluation of an experienced speech-language pathologist (SLP). Current approaches are insufficient for patient's needs, as one representative study described: "Patients rated 40% of the communication sessions with nurses as somewhat difficult to extremely difficult. Assistive communication strategies were uncommon, with little to no use of assistive communication materials (e.g., writing supplies, alphabet or word boards)." Designing an effective mode of communication for ICU patients unable to speak due to mechanical ventilation will likely improve patient's experiences and, potentially, long-term outcomes.

Some limited technologies exist to address these issues; however, they are not in widespread use due to a variety of reasons, including cost, lack of intuitiveness, and design that is not appropriate for the ICU setting. The investigators are designing a technological solution to assist ICU subjects in communicating with their caregivers, particularly nurses. The investigators are planning to do the initial testing of MOCS in the adult ICUs at the UMass Medical Center or at MGH.

The purpose of this stage of the project is to determine whether the device that has been designed in the previous study will be suitable for the needs of patients, families, and nurses. The investigators will be measuring duration of use, frequency and type of engagement, and mechanical stability.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are awake with a Glasgow Coma Scale score >10 (Motor 6, Verbal 0-1 [T], Eye opening 4) adult subjects at UMass Medical Center (Memorial and University ICUs) or at MGH (Bigelow 13, Lunder 6, Blake 7, Blake 12, or Ellison 4) are eligible for this study.
2. Both subjects who are able to speak and subjects who are unable to speak (due to intubation or tracheostomy) will be sought to be included in the study, although the focus will be on subjects who are unable to speak. (If additional feedback about the system from subjects who can speak would be helpful, this type of subject may be enrolled.)
3. Eligible subjects must have a history of being able to understand and communicate in written and spoken English, since the device software is in English.
4. May enroll both adults capable of consent and cognitively impaired adults, who will provide assent, if possible, and will have consent given by their legally authorized representative.

Exclusion Criteria:

1. non-adult individuals
2. prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Ability to use make selections in software using handheld component | 1 hour
  Able to make selection by squeezing handheld component, activating tablet software response, 5 times within 5 minutes of use (including training)

SECONDARY OUTCOMES:
Satisfaction assessed by modified SUS | 30 days
  Patients, nurses, and family members will be asked to indicate their level of satisfaction with the communication software using a homegrown instrument to assess usability (modeled partly on the System Usability Scale, or SUS). Four questions are derived from the SUS; they assess likelihood of recommending, ease of use, ease of learning, and perceived ability to use the system for communication. Each of these questions are assessed on a 1-5 scale, with higher values representing a better outcome. The subscales of these questions are averaged to reach a total score.
Duration of use | 1 hour
  The time spent using the system will be measured.
Level of engagement | 1 hour
  The number of each type of interaction with the system will be tabulated

CONTACTS AND LOCATIONS:
Overall Officials: J. Matthias Walz, MD, Principal Investigator — UMass Medical School
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - UMass Medical School, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No